CLINICAL TRIAL: NCT03597269
Title: Evaluation of Pneumococcal Vaccine Coverage
Acronym: SAUVAC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SAUVAC
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Immunocompromised Patients and Non-immunosuppressed Patients at Risk With an Indication for Pneumococcal Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumococcal infections are frequent and serious. Streptococcus pneumoniae is the leading cause of community-acquired pneumonia in adults. In metropolitan France, there are 6000 to 7000 bacteremic pneumococcal infections each year, with a mortality rate of 10 to 30% in adults.

To fight against these bacterial infections, vaccines have been developed. At a time when antibiotic savings and the fight against antimicrobial resistance are major public health issues, vaccination is a first choice option to slow the development of pneumococcal resistance. Thus, after these different actions, the proportions of pneumococci with decreased susceptibility to penicillin G fell from 53 to 22%.

While there is a significant decrease in invasive pneumococcal disease in children since the use of conjugate vaccines (vaccination of up to 94% of children), the rate of invasive Pneumococcal disease in adults has decreased less significantly.

In March 2017, the High Council of Public Health (HCSP) proposed the vaccination of all non-immunocompromised adults at risk and immunocompromised patients.

Awareness-raising among vaccinating physicians seems essential, especially in recent years when the value of vaccination is threatened by speculation about its efficacy and toxicity. However, the investigators know that vaccination aims not only to protect the individual, but also the population, especially children and the elderly and the fragile people.

Thus, in the context of pneumococcal vaccination, identifying one or more profiles of patients at risk in the absence of vaccination could be particularly beneficial. Indeed, if the physician knows about the population at risk of not being vaccinated, it will be better able to identify patients at risk of not being protected against pneumococcus.

ELIGIBILITY:
Inclusion Criteria:

* patient over the age of 18
* Patient without cognitive impairment
* Follow-up at the time of inclusion by a physician
* Patient with one or more indications for an anti-pneumococcal vaccination according to the 2017 vaccine recommendations
* Non-immunocompromised patients at risk, with underlying disease predisposing to the occurrence of invasive pneumococcal disease

Exclusion Criteria:

* Patient's opposition to participate
* Patients with the following contraindications to pneumococcal vaccination: severe acute infection in progress, allergy to one of the components vaccin
* Patient deprived of liberty
* Patient under guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population of the study corresponds to the patients who consulted in an emergency service in Paris during 3 months to determine the anti-pneumococcal vaccination coverage in adults at the scale of a Paris emergency service.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of Pneumococcal Vaccine Coverage in Adults with Pneumococcal Vaccine Indication | Day 1
  The primary outcome measure is to evaluate the patient's Immunization status for mandatory vaccinations, his pneumococcal vaccination status and how it was determined (the patient knew it, the presence of a vaccination card, attending physician, indeterminate status).

CONTACTS AND LOCATIONS:
Overall Officials: Cécile P CAISSO, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France